CLINICAL TRIAL: NCT00145158
Title: Phase I/II Study of Immunization With Multiple Peptides Mixed With the Immunological Adjuvant CpG 7909 or Montanide ISA51 in HLA-A2 Patients With Metastatic Cutaneous Melanoma
Brief Title: Immunization With 8 Peptides Mixed With CpG 7909 or Montanide ISA51 in Patients With Metastatic Cutaneous Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Availability of Investigational agent
Sponsor: Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2003-007
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Vaccine; Peptide; Montanide
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51; ProMune

STUDY DESIGN:
Intervention Model Description: The protocol planned the inclusion of 2 cohorts, each of them including 14 patients, with metastatic cutaneous melanoma, with at least one detectable metastasis (grades AJCC 2002 III N2b to N3, grades IV M1a, M1b, and M1c without elevation of the LDH rate and without central nervous system toxicity).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: 8 HLA-A2-restricted peptides and CpG 7909 (Experimental): Patients were immunized with a combination of 8 peptides corresponding to defined tumor antigens (MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2, NY-ESO-1.A2, NA17.A2 and Tyrosinase.A2), mixed with CpG 7909. Patients received six sequential injections at 2-week intervals.
  Interventions: Biological: 8 HLA-A2-restricted peptides and CpG 7909
- Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51 (Experimental): Patients were immunized with a combination of 8 peptides corresponding to defined tumor antigens (MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2, NY-ESO-1.A2, and NA17.A2), mixed with Montanide ISA 51. Tyrosinase.A2 was administered without Montanide ISA51. Patients received six sequential injections at 2-week intervals.
  Interventions: Biological: 8 HLA-A2-restricted peptides and Montanide ISA51

INTERVENTIONS:
Biological: 8 HLA-A2-restricted peptides and Montanide ISA51
  Arms: Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
Biological: 8 HLA-A2-restricted peptides and CpG 7909
  Arms: Cohort 1: 8 HLA-A2-restricted peptides and CpG 7909

SUMMARY:
The purposes of this study are to describe the immune response to individual peptides after immunization with a combination of 8 peptides and CpG 7909 or Montanide ISA51; to determine the safety of the vaccines and; to document the tumor response in patients receiving the vaccines.

DETAILED DESCRIPTION:
Patients received six sequential immunizations with 8 peptides presented by HLA-A2 and mixed with either CpG 7909 or Montanide ISA51, at 2-week intervals. The 8 peptides were injected at 8 distinct injection sites. These peptides are the following: MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2 (ALKD), and NA17.A2 (20% intradermally and 80% subcutaneously); NY-ESO-1.A2 and Tyrosinase.A2 (100% subcutaneously).

300 µg of each peptide (except MAGE-10.A2 150 µg) was mixed with 4 mg CpG 7909 (Cohort 1) or 0.5ml of Montanide ISA51 (Cohort 2). In Cohort 2, the Tyrosinase.A2 was administered without Montanide ISA51.

Tumor staging was performed before inclusion and at week 13. Peripheral Blood Lymphocytes (PBL) collections were performed before starting the treatment, and at weeks 3, 7 and 13. They provided the T lymphocytes for the immunological analysis.

At week 13, the PCR results of the pre-immune tumor biopsy must be available. Additional cycles of immunization, ONLY with the peptides expressed by the tumor, mixed with Montanide ISA51, will be proposed to patients without tumor progression requiring another treatment. A second cycle of 3 injections at 6-week intervals will be started at week 17, followed by a third cycle of 12 injections at 3-month intervals, starting at month 11. At any time, progression of the disease necessitating any treatment not allowed during the study will result in withdrawal.

The immune response may well be a limiting factor to the therapeutic efficacy of the vaccine. If this is the case, it then becomes crucial to understand why some patients develop a cytotoxic t-lymphocyte (CTL) response against the vaccine, while the majority of them do not. One possible explanation for the low frequency of clinical responses is that each injection of a single peptide has a low probability to provide the adequate stimulus to activate very rare CTL precursors. This probability should be increased if several peptides known to be undoubtedly associated with tumor regressions were used together to immunize patients.

ELIGIBILITY:
Inclusion Criteria

1. Histologically proven cutaneous melanoma, or clear cell sarcoma, which is considered as a subtype of melanoma.
2. Melanoma must be at one of the following AJCC 2002 stages:

   * Regional metastatic disease (any T; N2b, N2c or N3; M0).
   * Distant metastatic disease (any T; any N; M1a, M1b or M1c), except brain or leptomeningeal localizations, and except elevated LDH.
3. Patients must be HLA-A2.
4. A pre-immune tumor biopsy must be kept frozen for post-study PCR analysis.
5. Presence of at least one measurable or non-measurable tumor lesion.
6. Expected survival of at least 3 months.
7. Karnofsky performance scale ≥70 or WHO performance status of 0 or 1.
8. Within the last 4 weeks prior to study day 1, vital laboratory parameters should be within normal range, except for the following laboratory parameters, which must be within the ranges specified:

   Lab Parameter Range
   * Hemoglobin ≥ 10 g/dl or ≥ 6,25 mmol/l
   * Granulocytes ≥ 1,500/µl
   * Lymphocytes ≥ 700/µl
   * Platelets ≥ 100,000/µl
   * Serum creatinine ≤ 2.0 mg/dl or ≤ 177 μmol/l
   * Serum bilirubin ≤ 2.0 mg/dl or ≤ 34.2 μmol/l
   * ASAT and ALAT ≤ 2 x the normal upper limits
   * LDH ≤ the normal upper limit.
9. Viral tests:

   * HIV (human immunodeficiency virus): negative antibodies.
   * HBV (hepatitis B virus): negative antigens; antibodies may be positive.
   * HCV (hepatitis C virus): negative antibodies.
10. Age ≥ 18 years.
11. Able and willing to give valid written informed consent.

Exclusion Criteria

1. Previous treatment with more than one regimen of systemic chemotherapy, combined or not with non-specific immunotherapy such as interferon alpha or interleukins. Chemoimmunotherapy or radiotherapy must be stopped within the preceding 4 weeks (6 weeks for nitrosoureas and mitomycin C).
2. Clinically significant heart disease (NYHA Class III or IV) i.e. NYHA class 3 congestive heart failure; myocardial infarction within the past six months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias.
3. Active immunodeficiency or autoimmune disease. Vitiligo was not an exclusion criterion.
4. Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders, or other conditions requiring concurrent medications not allowed during this study.
5. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
6. Lack of availability for immunological and clinical follow-up assessments.
7. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
8. Pregnancy or breastfeeding.
9. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2007-11-30 (Actual); Study Completion 2009-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas VanBaren, MD, Study Chair — Ludwig Institute for Cancer Research; Thierry BOON, PhD, Study Director — Ludwig Institute for Cancer Research
Locations (2):
- Belgium (2):
  - Clinique Universitaires St-Luc, Brussels
  - Ludwig Institute for Cancer Research, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchand M, van Baren N, Weynants P, Brichard V, Dreno B, Tessier MH, Rankin E, Parmiani G, Arienti F, Humblet Y, Bourlond A, Vanwijck R, Lienard D, Beauduin M, Dietrich PY, Russo V, Kerger J, Masucci G, Jager E, De Greve J, Atzpodien J, Brasseur F, Coulie PG, van der Bruggen P, Boon T. Tumor regressions observed in patients with metastatic melanoma treated with an antigenic peptide encoded by gene MAGE-3 and presented by HLA-A1. Int J Cancer. 1999 Jan 18;80(2):219-30. doi: 10.1002/(sici)1097-0215(19990118)80:23.0.co;2-s. PMID 9935203
- [Background] Germeau C, Ma W, Schiavetti F, Lurquin C, Henry E, Vigneron N, Brasseur F, Lethe B, De Plaen E, Velu T, Boon T, Coulie PG. High frequency of antitumor T cells in the blood of melanoma patients before and after vaccination with tumor antigens. J Exp Med. 2005 Jan 17;201(2):241-8. doi: 10.1084/jem.20041379. PMID 15657293
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was to recruit 28 patients; 14 in each group. The first subject was treated on January 18, 2005. The study was prematurely closed in November 2007 as 6 of the 8 peptides had expired.
Groups:
- Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909: Patients with metastatic cutaneous melanoma, with at least one detectable metastasis (grades AJCC 2002 III N2b to N3, grades IV M1a, M1b, and M1c without elevation of the LDH rate and without central nervous system toxicity) received six sequential immunizations with 8 peptides presented by HLA-A2 and mixed with CpG 7909, at 2-week intervals. The 8 peptides were to be injected at 8 distinct injection sites. These peptides are the following: MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2 (ALKD), and NA17.A2 (20% intradermally and 80% subcutaneously); NY-ESO-1.A2 and Tyrosinase.A2 (100% subcutaneously).
- Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51: Patients with metastatic cutaneous melanoma, with at least one detectable metastasis (grades AJCC 2002 III N2b to N3, grades IV M1a, M1b, and M1c without elevation of the LDH rate and without central nervous system toxicity) received six sequential immunizations with 8 peptides presented by HLA-A2 and mixed with Montanide ISA51, at 2-week intervals. The 8 peptides were to be injected at 8 distinct injection sites. These peptides are the following: MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2 (ALKD), and NA17.A2 (20% intradermally and 80% subcutaneously); NY-ESO-1.A2 and Tyrosinase.A2 (100% subcutaneously). The Tyrosinase.A2 was administered without Montanide ISA51.
Period: Overall Study
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
Started | 16 | 7
Completed | 14 | 4
Not Completed | 2 | 3
Not completed — premature withdrawal | 2 | 3

BASELINE CHARACTERISTICS:
Population: All patients who received at least one immunization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51 | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Customized [Count of Participants; unit: Participants]
  ≥ to 18 years | 16 | 7 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  Belgium | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Cytotoxic T-lymphocyte (CTL) Response to Individual Peptides After Immunization With a Combination of 8 Peptides and CpG 7909 or Montanide ISA51.
Description: Peripheral blood lymphocytes (PBL) were collected prior to the first dose of vaccine and after the completion of the six vaccinations in Week 13. Specific CTL directed against the 8 vaccine antigens ( NA17.A2, MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2 and Tyrosinase.A2) was assessed by using re-stimulation in vitro, followed by staining with the corresponding tetramer (MLPC/tetramer). A patient was considered to have a positive CTL response when the post-vaccine CTL response against at least one of the vaccine antigens was ten times higher than the corresponding pre-treatment value.
Time Frame: Week 13
Population: Patients who received at least six vaccinations and had samples taken at Week 13.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
Number analyzed (Participants) | 14 | 3
Participants
  Patients with CTL Response | 6 | 1
  Patients with no CTL Response | 8 | 2

2. Secondary Outcome: Number of Patients With Dose Limiting Toxicities (DLT).
Description: Toxicity was evaluated according to the National Cancer Institute (CTC Scale Version 3.0, published December 12, 2003).
  Dose limiting toxicity (DLT) is defined as:
  * Any Grade 3 hematological or non-hematological toxicity other than skin or flu-like symptoms
  * Any Grade 4 toxicity To be dose-limiting, an adverse event must be definitely, probably, or possibly related to the administration of the investigational agent.
Time Frame: up to Week 13
Population: All patients who received at least one immunization.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
Number analyzed (Participants) | 16 | 7
Participants | 2 | 0

3. Secondary Outcome: Number of Patients With Tumor Responses After Immunization With a Combination of 8 Peptides and CpG 7909 or Montanide ISA51 as Measured by RECIST.
Description: Tumor response was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST). Tumor measurements were taken at screening and at the end of Cycle 1 in Week 13. Per RECIST, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Week 13
Population: Patients who received at least six immunizations and had tumor response measured at Week 13.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909: Patients with metastatic cutaneous melanoma, with at least one detectable metastasis (grades AJCC 2002 III N2b to N3, grades IV M1a, M1b, and M1c without elevation of the LDH rate and without central nervous system toxicity) received six sequential immunizations with 8 peptides presented by HLA-A2 and mixed with CpG 7909, at 2-week intervals. The 8 peptides were injected at 8 distinct injection sites. These peptides are the following: MAGE-1.A2, MAGE-3.A2, MAGE-4.A2, MAGE-10.A2, MAGE-C2.A2 (ALKD), and NA17.A2 (20% intradermally and 80% subcutaneously); NY-ESO-1.A2 and Tyrosinase.A2 (100% subcutaneously).
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
Number analyzed (Participants) | 14 | 4
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 4 | 0
  Progressive Disease (PD) | 10 | 4

4. Secondary Outcome: Number of Patients With Cytotoxic T-lymphocyte (CTL) Responses and Tumor Expression of the Corresponding Genes.
Description: Gene expression was determined by RT-PCR on a pre-treatment tumor sample. The correlation of the induction of a CTL response against a defined antigen to the prior expression of the gene coding for this antigen by the tumor removed before vaccination was assessed.
Time Frame: Week 13
Population: Patients who had pretreatment tumor samples analyzed for gene expression, received at least six immunizations and had CTL responses at Week 13.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
Number analyzed (Participants) | 6 | 1
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: up to 45 months
Description: All adverse events (AEs) occurring during the study were to be documented in the source records and on the respective AE Case Report Form (CRF), regardless of the assumption of a causal relationship. All events, which occurred after signed informed consent, were to be documented. Toxicities were graded according to the scale of the National Cancer Institute, CTC Scale Version 3.0, published on December 12, 2003.
Arm/Group | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 7/16 | 3/7
Other Adverse Events (participants affected / at risk) | 16/16 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 (N=16) | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51 (N=7)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 8 HLA-A2-restricted Peptides and CpG 7909 (N=16) | Cohort 2: 8 HLA-A2-Restricted Peptides and Montanide ISA51 (N=7)
Injection site erythema (General disorders) | 16 | 6
Injection site pain (General disorders) | 14 | 2
Injection site induration (General disorders) | 11 | 2
Fatigue (General disorders) | 8 | 3
Pyrexia (General disorders) | 9 | 1
Injection site warmth (General disorders) | 8 | 1
Influenza like illness (General disorders) | 6 | 0
Injection site pruritus (General disorders) | 4 | 2
Asthenia (General disorders) | 5 | 0
Malaise (General disorders) | 4 | 1
Injection site oedema (General disorders) | 3 | 1
Injection site swelling (General disorders) | 2 | 2
Injection site reaction (General disorders) | 1 | 2
Injection site ulcer (General disorders) | 3 | 0
Axillary pain (General disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Nodule (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Illness (General disorders) | 1 | 0
Injection site erosion (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 0 | 1
Injection site joint pain (General disorders) | 1 | 0
Injection site scab (General disorders) | 1 | 0
Injection site vesicles (General disorders) | 1 | 0
Mass (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0
General physical condition abnormal (Investigations) | 6 | 0
Weight decreased (Investigations) | 4 | 2
Respiratory rate increased (Investigations) | 3 | 1
Antinuclear antibody positive (Investigations) | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Karnofsky scale worsened (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Inflammatory marker increased (Investigations) | 1 | 0
Karnofsky scale (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Tumor ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Depression (Psychiatric disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depressed mood (Psychiatric disorders) | 0 | 2
Nervousness (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Scrotal infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 4 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysstasia (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Heamorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No